CLINICAL TRIAL: NCT01263327
Title: An Open-Label, Single-dose, Non-Randomized, Safety and Tolerability Study of Recombinant Human Papillomavirus Virus 16/18 Bivalent Vaccine (E.Coli)in Healthy Female Subjects Aged 18 to 55 Years
Brief Title: Clinical Trial of Recombinant Human Papillomavirus Virus 16/18 Bivalent Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xiamen University (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Zhang, Professor, Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HPV-PRO-001
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Cervical Cancer
Keywords: human papillomavirus vaccine
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HPV 16/18 (Experimental): Participants in this arm would intramuscularly receive 90mcg of HPV 16/18 bivalent vaccine at 0, 1, 6 month for 3 doses.
  Interventions: Biological: HPV 16/18

INTERVENTIONS:
Biological: HPV 16/18 — Participants would intramuscularly receive 90mcg of HPV 16/18 bivalent vaccine at 0, 1, 6 month for 3 doses.

SUMMARY:
This phase I clinical study was designed to evaluate the safety of novel recombinant HPV 16/18 bivalent vaccine, manufactured by Xiamen Innovax Biotech CO., LTD., in healthy women 18-55 years of age at enrolment. Approximately 30 study subjects will receive the novel HPV vaccine administered intramuscularly according to a 0-1-6 month schedule.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the subject prior to enrolment;
* Female between, and including, 18 and 55 years of age at the time of enrolment;
* Subjects must be free of obvious health problems;
* Not pregnant and having no plan for pregnancy;

Exclusion Criteria:

* Pregnant or breastfeeding or having plan for pregnancy during the whole study (Month 0-7);
* Previous vaccination against HPV;
* Having severe allergic history or other immunodeficiency;
* Chemotherapy and other immunosuppressive agents using;

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Measure injection-site complaints within 7 days after each vaccination; Measure systematic adverse reactions within 1 month after vaccination; Measure serious adverse experience; Measure blood, liver and kidney functions pre- and 3 days post vaccination. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Yue-mei Hu, Bachelor, Principal Investigator — Jiangsu Provincial Centre for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Centre for Disease Control and Prevention, Dongtai, Jiangsu, China

REFERENCES:
- [Result] Hu YM, Huang SJ, Chu K, Wu T, Wang ZZ, Yang CL, Cai JP, Jiang HM, Wang YJ, Guo M, Liu XH, Huang HJ, Zhu FC, Zhang J, Xia NS. Safety of an Escherichia coli-expressed bivalent human papillomavirus (types 16 and 18) L1 virus-like particle vaccine: an open-label phase I clinical trial. Hum Vaccin Immunother. 2014;10(2):469-75. doi: 10.4161/hv.26846. Epub 2013 Oct 25. PMID 24161937